CLINICAL TRIAL: NCT00673231
Title: A 24-week International, Randomized, Parallel-group, Double-blind, Placebo-controlled Phase III Study With a 80-week Extension Period to Evaluate the Efficacy and Safety of Dapagliflozin Therapy When Added to the Therapy of Patients With Type 2 Diabetes With Inadequate Glycaemic Control on Insulin
Brief Title: Efficacy and Safety of Dapagliflozin, Added to Therapy of Patients With Type 2 Diabetes With Inadequate Glycemic Control on Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00006
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes
Keywords: Dapagliflozin; efficacy; safety; add on to insulin; Oral AntiDiabetic; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 2.5mg
  Interventions: Drug: Dapagliflozin
- 2 (Experimental): 5mg
  Interventions: Drug: Dapagliflozin
- 3 (Experimental): 10mg
  Interventions: Drug: Dapagliflozin
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — tablet oral 2.5 mg total daily dose once daily 48 weeks (= 24 week randomised treatment period + 24 week study extension period I)
  Arms: 1
Drug: Dapagliflozin — Tablet oral 5 mg total daily dose once daily 48 weeks (= 24 week randomised treatment period + 24 week study extension period I)
  Arms: 2
Drug: Dapagliflozin — Tablet oral 10 mg total daily dose once daily 48 weeks (= 24 week randomised treatment period + 24 week study extension period I)
  Arms: 3
Drug: Placebo — Placebo
  Arms: 4
Drug: Dapagliflozin — tablet oral 2.5 total daily dose once daily 56 weeks (= 56 week study extension period II)
  Arms: 1
Drug: Dapagliflozin — tablet oral 10 mg total daily dose once daily 56 weeks (= 56 week study extension period II)patients that have been treated with 5 mg during the 24 week randomised treatment period and extension I period will during extension II period switched to 10 mg
  Arms: 3

SUMMARY:
This study is being carried out to see if Dapagliflozin in addition to insulin is effective and safe in treating patients with type 2 diabetes when compared to placebo (identical looking inactive treatment) in addition to insulin

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Patients with HbA1c ≥7.5% and ≤10.5% and who are on a stable insulin regimen of at least 30 IU of injectable insulin per day either without any other oral antidiabetic drug or with a stable dose of oral antidiabetic drugs

Exclusion Criteria:

* Type 1 Diabetes
* Treatment with more than two additional oral antidiabetic drugs
* Moderate and severe renal (kidney) failure or dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Wilding, MD, Principal Investigator — Clinical Sciences CentreUniversity Hospital AintreeLongmoor LaneLiverpool, UK
Locations (92):
- United States (13):
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, Roswell, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Omaha, Nebraska
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
- Austria (2):
  - Research Site, Salzburg
  - Research Site, Vienna
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (18):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Langley, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Etobicoke, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Mirabel, Quebec
  - Research Site, Sherbrooke, Quebec
- Finland (8):
  - Research Site, Lahti, Finland
  - Research Site, Helsinki
  - Research Site, Joensuu
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Seinäjoki
  - Research Site, Turku
- Germany (9):
  - Research Site, Bad Oeynhausen
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Magdeburg
  - Research Site, Münster
  - Research Site, Riesa
  - Research Site, Wolmirstedt
- Hungary (9):
  - Research Site, Csongrád
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Komárom
  - Research Site, Miskolc
  - Research Site, Székesfehérvár
  - Research Site, Veszprém
- Netherlands (4):
  - Research Site, Amersfoort
  - Research Site, Den Helder
  - Research Site, Leiden
  - Research Site, Rotterdam
- Romania (3):
  - Research Site, Brasov, Brașov County
  - Research Site, Tg Mures, Mureș County
  - Research Site, Bucharest
- Russia (3):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
- Slovakia (7):
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Považská Bystrica
  - Research Site, Prešov
- Spain (4):
  - Research Site, Seville, Andalusia
  - Research Site, Sabadell (barcelona), Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, Alicante, Valencia
- United Kingdom (8):
  - Research Site, Reading, Berks
  - Research Site, Aylesbury, Bucks
  - Research Site, Ashford
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Liverpool
  - Research Site, Reading
  - Research Site, Swansea

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Aberle J, Menzen M, Schmid SM, Terkamp C, Jaeckel E, Rohwedder K, Scheerer MF, Xu J, Tang W, Birkenfeld AL. Dapagliflozin effects on haematocrit, red blood cell count and reticulocytes in insulin-treated patients with type 2 diabetes. Sci Rep. 2020 Dec 28;10(1):22396. doi: 10.1038/s41598-020-78734-z. PMID 33372185
- [Derived] Shah M, Stolbov L, Yakovleva T, Tang W, Sokolov V, Penland RC, Boulton D, Parkinson J. A model-based approach to investigating the relationship between glucose-insulin dynamics and dapagliflozin treatment effect in patients with type 2 diabetes. Diabetes Obes Metab. 2021 Apr;23(4):991-1000. doi: 10.1111/dom.14305. Epub 2021 Jan 25. PMID 33368935
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- [Derived] van Haalen HG, Pompen M, Bergenheim K, McEwan P, Townsend R, Roudaut M. Cost effectiveness of adding dapagliflozin to insulin for the treatment of type 2 diabetes mellitus in the Netherlands. Clin Drug Investig. 2014 Feb;34(2):135-46. doi: 10.1007/s40261-013-0155-0. PMID 24243529
- [Derived] Wilding JP, Woo V, Rohwedder K, Sugg J, Parikh S; Dapagliflozin 006 Study Group. Dapagliflozin in patients with type 2 diabetes receiving high doses of insulin: efficacy and safety over 2 years. Diabetes Obes Metab. 2014 Feb;16(2):124-36. doi: 10.1111/dom.12187. Epub 2013 Aug 29. PMID 23911013
- [Derived] Wilding JP, Woo V, Soler NG, Pahor A, Sugg J, Rohwedder K, Parikh S; Studiengruppe Dapagliflozin 006. [Long-term efficacy of dapagliflozin in patients with type 2 diabetes mellitus receiving high doses of insulin]. Dtsch Med Wochenschr. 2013 Apr;138 Suppl 1:S27-38. doi: 10.1055/s-0032-1305284. Epub 2013 Mar 25. German. PMID 23529568
- [Derived] Wilding JP, Woo V, Soler NG, Pahor A, Sugg J, Rohwedder K, Parikh S; Dapagliflozin 006 Study Group. Long-term efficacy of dapagliflozin in patients with type 2 diabetes mellitus receiving high doses of insulin: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):405-15. doi: 10.7326/0003-4819-156-6-201203200-00003. PMID 22431673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 30 April 2008, Last participant completed 24 week period: 19 May 2009. 1240 enrolled at 126 centres in 13 countries. Men and women aged ≥18-≤80 years at time of consenting who have inadequate glycaemic control (HbA1c ≥7.5% and ≤10.5%) and are on a stable insulin regimen (≥30 IU of injectable insulin per day for 8 weeks).
Pre-assignment Details: For two weeks prior to randomization, participants recorded their daily self monitored plasma glucose and insulin use. At randomization, qualified participants were stratified according to their use of other anti-diabetic (OAD) medication or not. No more than 60% of enrolled participants were to take insulin plus OADs.
Groups:
- Dapagliflozin 2.5mg: Dapagliflozin tablet oral 2.5 mg total daily dose once daily 24 weeks
- Dapagliflozin 5mg: Dapagliflozin tablet oral 5 mg total daily dose once daily 24 weeks
- Dapagliflozin 10mg: Dapagliflozin tablet oral 10 mg total daily dose once daily 24 weeks
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Started | 197 (Of the 197 randomized participants only 193 were included in the full analysis set) | 202 (All 202 were included in the full analysis set) | 212 (Of the 212 randomized participants only 211 were included in the full analysis set) | 196 (Of the 196 randomized participants only 194 were included in the full analysis set)
Completed | 168 | 180 | 186 | 178
Not Completed | 29 | 22 | 26 | 18
Not completed — Withdrawal by Subject | 14 | 10 | 8 | 6
Not completed — Adverse Event | 6 | 5 | 9 | 6
Not completed — Lost to Follow-up | 1 | 2 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Study criteria,compliance,safety, other | 8 | 5 | 7 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg | Total
Number analyzed (Participants) | 193 | 202 | 211 | 194 | 800
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (8.61) | 59.8 (7.64) | 59.3 (7.91) | 59.3 (8.75) | 59.3 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 102 | 111 | 107 | 418
  Male | 95 | 100 | 100 | 87 | 382
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 186 | 190 | 200 | 184 | 760
  Black/African American | 6 | 3 | 5 | 5 | 19
  Asian | 0 | 7 | 3 | 3 | 13
  Other | 1 | 2 | 3 | 2 | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 33.14 (5.862) | 32.95 (5.032) | 32.97 (5.261) | 33.41 (5.061) | 33.11 (5.303)
HbA1C [Mean (Standard Deviation); unit: Percent] | 8.47 (0.768) | 8.46 (0.780) | 8.62 (0.892) | 8.57 (0.820) | 8.53 (0.819)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dl] | 170.62 (57.165) | 180.11 (59.9) | 185.38 (58.712) | 173.09 (54.916) | 177.58 (57.950)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To assess the efficacy of 2.5 mg, 5 mg and 10 mg dapagliflozin compared to placebo as add-on therapy to insulin in improving glycaemic control in participants with type 2 diabetes who have inadequate glycaemic control on ≥ 30 IU injectable insulin daily for at least 8 weeks prior to enrolment, as determined by the change in HbA1c levels from baseline to Week 24, excluding data after insulin up-titration.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Number analyzed (Participants) | 188 | 198 | 210 | 192
Percent | -0.30 [-0.40 to -0.20] | -0.75 [-0.85 to -0.65] | -0.82 [-0.92 to -0.73] | -0.90 [-1.00 to -0.80]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 2.5mg; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0 (with alpha = 0.019 applying Dunnett's adjustment, two-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.019 (2-sided) applying Dunnett's adjustment. A hierarchical closed testing procedure was used to control the Type I error rate across the primary and key secondary endpoints; with treatment group (all treatment groups included) and stratum (other oral anti-diabetic med use) as effect and baseline value as covariate; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.59 to -0.31], Standard Error of Mean 0.0726
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 5mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.66 to -0.38], Standard Error of Mean 0.0718
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 10mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.74 to -0.45], Standard Error of Mean 0.0733

2. Secondary Outcome: Adjusted Mean Change in Body Weight
Description: To examine whether treatment with dapagliflozin in combination with insulin is superior in reducing body weight or causing less weight gain as compared to placebo added to insulin treatment after 24 weeks of treatment (LOCF), excluding data after insulin up-titration.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Number analyzed (Participants) | 188 | 198 | 210 | 192
kg | 0.02 [-0.34 to 0.38] | -0.98 [-1.33 to -0.63] | -0.98 [-1.32 to -0.64] | -1.67 [-2.02 to -1.31]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 2.5mg; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0001, ANCOVA — significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure within treatment group; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.50 to -0.49], Standard Error of Mean 0.2560
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 5mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.50 to -0.50], Standard Error of Mean 0.2523
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 10mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-2.19 to -1.18], Standard Error of Mean 0.2578

3. Secondary Outcome: Adjusted Mean Change in Calculated Mean Daily Insulin Dose
Description: To examine whether treatment with dapagliflozin in combination with insulin leads to a lower absolute calculated mean daily insulin dose as compared to placebo added to insulin treatment alone, from baseline to week 24, including data after insulin up-titration.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: IU/day
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Number analyzed (Participants) | 191 | 200 | 209 | 194
IU/day | 5.08 [3.23 to 6.93] | -1.80 [-3.60 to 0.01] | -0.61 [-2.38 to 1.15] | -1.16 [-2.99 to 0.68]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 2.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.87, 95% CI 2-sided [-9.46 to -4.28], Standard Error of Mean 1.3195
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 5mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.69, 95% CI 2-sided [-8.25 to -3.13], Standard Error of Mean 1.3045
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 10mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.23, 95% CI 2-sided [-8.84 to -3.63], Standard Error of Mean 1.3286

4. Secondary Outcome: Proportion of Participants With Calculated Mean Daily Insulin Dose Reduction
Description: To examine whether treatment with dapagliflozin in combination with insulin leads to higher percentage of participants with calculated mean daily insulin dose reduction from baseline to week 24 (i.e. reduction >= 10%) as compared to placebo added to insulin treatment.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Number analyzed (Participants) | 191 | 200 | 209 | 194
Percentage of participants | 11.0 [6.5 to 15.4] | 18.1 [12.8 to 23.4] | 16.8 [11.7 to 21.8] | 19.7 [14.1 to 25.2]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 2.5mg; H0: proportion(treat) minus proportion(placebo) = 0 versus the alternative HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p = 0.0427, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, adjustment for stratum (other oral anti-diab med use) and baseline value; Risk Difference (RD) = 7.2, 95% CI 2-sided [0.2 to 14.1], Standard Error of Mean 3.536
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 5mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0903, Regression, Logistic — not significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure within treatment group; [statistical method as in outcome 4, analysis 1]; Risk Difference (RD) = 5.8, 95% CI 2-sided [-0.9 to 12.5], Standard Error of Mean 3.434
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 10mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0166, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 4, analysis 1]; Risk Difference (RD) = 8.7, 95% CI 2-sided [1.6 to 15.8], Standard Error of Mean 3.634

5. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose (FPG)
Description: To examine whether treatment with dapagliflozin in combination with insulin is superior in reducing Fasting Plasma Glucose (FPG) as compared to placebo added to insulin treatment after 24 weeks of treatment, excluding data after insulin up-titration.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Number analyzed (Participants) | 177 | 190 | 204 | 183
mg/dL | 3.3 [-3.3 to 9.9] | -12.5 [-18.9 to -6.1] | -18.8 [-25.0 to -12.7] | -21.7 [-28.2 to -15.2]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 2.5mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -15.8, 95% CI 2-sided [-25.0 to -6.6], Standard Error of Mean 4.684
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 5mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANCOVA — Not significant. Hierarchical closed testing procedure within treatment group stopped at previous endpoint; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -22.1, 95% CI 2-sided [-31.2 to -13.1], Standard Error of Mean 4.616
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 10mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -25.0, 95% CI 2-sided [-34.3 to -15.8], Standard Error of Mean 4.718

6. Other Pre Specified Outcome: Proportion of Participants With Lack of Glycemic Control
Description: Participants with lack of glycemic control or insulin up-titration for failing to achieve pre-specified glycemic targets
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Number analyzed (Participants) | 193 | 202 | 211 | 194
Participants | 54 | 22 | 24 | 19

ADVERSE EVENTS:
Time Frame: Non-serious/serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment period plus 4/30 days or up to follow-up visit if earlier, or up to and incl the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Placebo | Dapagliflozin 2.5mg | Dapagliflozin 5mg | Dapagliflozin 10mg
Serious Adverse Events (participants affected / at risk) | 14/197 | 15/202 | 10/212 | 14/196
Other Adverse Events (participants affected / at risk) | 115/197 | 135/202 | 128/212 | 107/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=197) | Dapagliflozin 2.5mg (N=202) | Dapagliflozin 5mg (N=212) | Dapagliflozin 10mg (N=196)
Angina Pectoris (Cardiac disorders) | 0 | 1 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 0 | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 2 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Change Of Bowel Habit (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Dislocation Of Joint Prosthesis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thrombosis In Device (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 2 | 0 | 0 | 0
Burning Sensation (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid Artery Occlusion (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1 | 0 | 1
Hypoglycaemic Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Aortic Valve Replacement (Surgical and medical procedures) | 0 | 0 | 1 | 0
Diabetic Microangiopathy (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=197) | Dapagliflozin 2.5mg (N=202) | Dapagliflozin 5mg (N=212) | Dapagliflozin 10mg (N=196)
Nasopharyngitis (Infections and infestations) | 22 | 28 | 29 | 17
Urinary Tract Infection (Infections and infestations) | 6 | 10 | 12 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 5 | 6 | 6
Headache (Nervous system disorders) | 14 | 8 | 9 | 2
Hypertension (Vascular disorders) | 16 | 11 | 13 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 8 | 4 | 9
Hypoglycemia (Endocrine disorders) | 83 | 111 | 101 | 88

LIMITATIONS AND CAVEATS:
For participants who did not complete 24 weeks LOCF (last observation carried forward) was used. Only values prior to insulin up-titration were used for outcome measures except for mean daily insulin dose which was evaluated regardless of.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.